CLINICAL TRIAL: NCT04921930
Title: Evaluation of the Effect of Artesunate in Friedreich Ataxia (FA) Phase I-II Efficacy-Toxicity of Artesunate in Friedreich Ataxia
Brief Title: Evaluation of the Effect of Artesunate in Friedreich Ataxia (FA)
Acronym: ARTEMIS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Imagine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C20-54
Record Dates: First submitted 2021-05-31; First posted 2021-06-10 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Artesunate (Experimental): Dose escalation of oral artesunate:
  Step 1: 25 mg daily (1 tablet) during one week Step 2: 50 mg daily (2 tablets) during one week (if no effect on biomarker and no adverse reaction at step 1) Step 3: 75 mg daily (3 tablets) during one week (if no effect on biomarker and no adverse reaction at step 2) Step 4: 100 mg daily (4 tablets) duing one week (if no efficacy and no adverse reaction at step 3)
  Interventions: Drug: Artesunate Oral Product

INTERVENTIONS:
Drug: Artesunate Oral Product — Dose escalation intake of artesunate

SUMMARY:
This dose-escalation study is aimed at investigating a novel application for artesunate in the treatment of Friedreich ataxia. It will evaluate this novel application of oral artesunate using a surrogate biological marker as primary endpoint in a phase I-II open trial

ELIGIBILITY:
Inclusion Criteria:

* Patients with FA confirmed by genetic analysis
* Weight of at least 50 kg
* Compliant patient agreeing to come to all protocol visits
* Signature of consent form by patient or parents of minor patient
* Patients with no treatment during 30 days prior to the first intake of study drug, except cardiac, diabetes and spasticity treatments
* Patients agreeing to use effective contraception for the duration of the study and up to 91 days after the last dose of the study treatment
* Affiliation to an Health Insurance Scheme of beneficiary of such a scheme

Exclusion Criteria:

* Patient under justice protection
* Female patients
* Abnormal biological values of renal and liver functions and cell blood count (CBC)
* Progressive associated disease
* Treatment interfering with iron transport within 30 days before first intake of artesunate
* Participation to another clinical trial
* Hypersensitivity to artesunate or to any component of the drug
* Blood potassium lower than normal value
* QT / QTc interval > 450 ms on the ECG performed at inclusion
* Congenital long QT syndrome
* Family history of sudden cardiac death before the age of 50
* Heart disease: ischemia or myocardial infarction, congestive heart failure or conduction disorder in the 6 months preceding inclusion
* History of arrhythmia
* Electrolyte imbalances: hypomagnesemia, hypocalcemia
* Bradycardia (<50 beats per minute)
* Acute neurological events within 6 months prior to inclusion

Ages: 16 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Search for the maximal tolerated and effective dose of oral artesunate to regulate iron homeostasis and Transferrin 1 receptor (TfR1) immunofluorescence in Peripheral Blood Mononuclear Cells (PBMCs) | at Day 7 (last day of drug intake)
  Evaluation of the biological efficacy on an ex vivo marker in the absence of observed side effects. This is a binary criterion established by comparison between compared measurements of the biomarker. If an effect on the biomarker is observed from the initial dose, the dose escalation will stop as the "ex-vivo" efficacy criterion is met. Otherwise the test will be repeated at an escalating dose. If an adverse effect is observed for a given dose, the maximal tolerated dose will be considered to be the immediately lower dose.

SECONDARY OUTCOMES:
Incidence of Adverse Events with Artesunate in FA patients | From first intake to 30 days after last intake of study drug
  Rate of side effects according artesunate doses
Type of Adverse Events with Artesunate in FA patients | From first intake to 30 days after last intake of study drug
  Desciption of side effects according artesunate doses
Impact of stopping an effective dose of artesunate on the regulation of iron homeostasis and TfR1 immunofluorescence | At Day 14 (7 days after the last drug intake)
  Evolution of the response to treatment after one week without treatment in patients who presented a positive response: Comparison of the results of intracellular iron concentration in in vitro PBMCs obtained with the sample at the end of the week without treatment with those obtained at the end of the week under treatment at a given dose

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Munnich, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Centre d'Investigation Clinique, hôpital Necker Enfants Malades, Paris, France